CLINICAL TRIAL: NCT01013571
Title: A Canadian, Phase IV, Multicenter, Comparative, Open-label Study Evaluating 2 Approaches of Blood Glucose Monitoring and Insulin Titration (Patient-managed vs Health Care Professional) in T2DM Patients While Receiving the Addition of 1 Injection of Insulin Glulisine at Breakfast Following Optimization of Insulin Glargine
Brief Title: Self Titration With Apidra to Reach Target Study (START)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_04695
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine

ARMS (2):
- 1 (Experimental): 12-week run-in phase with Glargine +/- OADs followed by 24-week treatment phase with glulisine (AM) + glargine ; health care professional-managed
  Interventions: Drug: insulin glargine; Drug: Apidra (insulin glulisine)
- 2 (Experimental): 12-week run-in phase with Glargine +/- OADs followed by 24-week treatment phase with glulisine (AM) + glargine ; patient-managed
  Interventions: Drug: insulin glargine; Drug: Apidra (insulin glulisine)

INTERVENTIONS:
Drug: insulin glargine — pre-filled disposable pen, in package of 5.
Drug: Apidra (insulin glulisine) — pre-filled disposable pen, in package of 5

SUMMARY:
Primary Objective:

The primary objective of this study is to demonstrate non-inferiority of a patient-managed titration algorithm (including blood glucose monitoring) for the addition of a single dose of insulin glulisine at breakfast in Canadian patients with inadequately controlled T2DM after optimization of basal insulin, compared with an HCP-managed titration algorithm. The primary endpoint for assessment of this objective is the percent of patients reaching a target HbA1c <=7.0% without severe hypoglycemia at the end of the study.

Secondary Objective:

Secondary objectives of the study are to compare the effect of the two different insulin glulisine titration algorithms (patient-managed versus HCP-managed) on the following:

* change in HbA1c, FG, and 7-point glucose profile at Week 24 and Week 36
* satisfaction with treatment (DTSQc for patient and questionnaire for HCP) at Week 36
* change in weight at Week 24 and Week 36
* incidence of hypoglycemia
* insulin doses
* resource utilization (rural/urban, blood glucose meter test strips, lancets, HCP visits, telephone calls, and hospitalizations)
* adherence with the patient-managed monitoring algorithm

ELIGIBILITY:
Inclusion criteria:

Run-in phase:

* T2DM
* Treated for at least 3 months with a basal insulin (insulin glargine, NPH, detemir) +/- oral antidiabetic drugs (OADs) with an HbA1c >7.0% or insulin naive (2-3 OADs) with an HbA1c >=7.8% (historic HbA1c result up to 3 months of screening is acceptable)

Randomized treatment phase:

* Completed run-in phase
* HbA1c >7.0% and >= 1 episode of confirmed nocturnal hypoglycemia (BG <4.0 mmol/L) or >= 2 measurements of FG <=6.0 mmol/L within the previous week Patients who completed the run-in phase with HbA1c >7.0% and did not meet the randomization criteria will continue titrating insulin glargine and be followed until the end of study.

Exclusion Criteria:

* No food intake before lunch (noon)
* Unstable diet intake or significant changes to current diet regimen
* Nightshift worker
* Type 1 Diabetes Mellitus
* Subjects unwilling to inject insulin or perform self-monitoring blood glucose
* Pregnant, alcohol or drug abuse
* Active cancer or any other disease or condition which in the opinion of the investigator would make the subject unsuitable for participation in the study
* Any clinical significant laboratory findings that in the judgment of the investigator would preclude safe completion of the study
* Known allergies to study drugs

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects reaching target HbA1c <=7.0% without severe hypoglycemia | at week 36 (end of study)

SECONDARY OUTCOMES:
Change in HbA1c, FG, and 7-point glucose profile | from Week 12 (randomization) to Week 24 and Week 36
Change in weight | from Week 12 to Week 24 and to Week 36
Incidence of hypoglycemia | Week 12 , Week 24 and Week 36
Treatment satisfaction (DTSQ for patient ) | from Week 12 to Week 36
Adherence with the patient-managed monitoring algorithm | Week 12 , Week 24 and Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Laval, Canada

REFERENCES:
- [Derived] Harris SB, Yale JF, Berard L, Stewart J, Abbaszadeh B, Webster-Bogaert S, Gerstein HC. Does a patient-managed insulin intensification strategy with insulin glargine and insulin glulisine provide similar glycemic control as a physician-managed strategy? Results of the START (Self-Titration With Apidra to Reach Target) Study: a randomized noninferiority trial. Diabetes Care. 2014;37(3):604-10. doi: 10.2337/dc13-1636. Epub 2013 Oct 29. PMID 24170757